CLINICAL TRIAL: NCT00798538
Title: Integration of Buprenorphine Into HIV Clinical Settings - Primary Care Model (PCM)
Acronym: BELIEVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Waterbury Hospital (Unknown); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); The New York Academy of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H97HA03800-03
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Buprenorphine; HIV; Drug Abuse; Drug Addiction; Drug Dependence; Drug Use Disorders; Drug Use Disorder; Substance Abuse; Opiate Addiction; Substance-related Disorders
Keywords: Buprenorphine; HIV; Drug Abuse; Drug Addiction; Drug Dependence; Drug Use Disorders; Drug Use Disorder; Substance Abuse; Opiate Addiction; Substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated (Active Comparator): Provision of buprenorphine induction and management, substance abuse counseling and HIV care at one clinic.
  Interventions: Other: Services will be provided at one site
- Non-integrated (Placebo Comparator): Buprenorphine induction, substance abuse counseling and HIV care will be managed at multiple locations, respectively: the Community Health Care Van, the Yale AIDS Program, and individuals' HIV clinics.
  Interventions: Other: Services remain dispersed; i.e., not centralized to one-location or provider.

INTERVENTIONS:
Other: Services will be provided at one site — Provision of buprenorphine induction and management, substance abuse counseling and HIV care will be provided at one clinic: the Waterbury Hospital Infectious Disease Clinic..
  Arms: Integrated
Other: Services remain dispersed; i.e., not centralized to one-location or provider. — Buprenorphine induction, substance abuse counseling, and HIV care will be provided at separate locations: the Community Health Care Van (CHCV), the Yale AIDS Program, and patients' own HIV providers, respectively.
  Arms: Non-integrated

SUMMARY:
The purpose of this study is to assess the feasibility, cost and effectiveness of interventions designed to integrate buprenorphine treatment for opioid dependence into HIV primary care in ten HIV care centers in the U.S.

In the site led by Dr. Altice, we compare two models of providing HIV care and buprenorphine treatment. Assignments are based on participants' city of residence. In the onsite (integrated care) model, participants receive buprenorphine, substance abuse counseling and HIV care at one location: the Waterbury Hospital Infectious Disease Clinic. In the off-site model (non-integrated care) buprenorphine induction, substance abuse counseling, and HIV care will be provided at separate locations: the Community Health Care Van (CHCV), the Yale AIDS Program, and patients' own HIV providers, respectively. Data is collected from interviews with participants, reviews of medical records, and surveys and interviews with clinicians.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Clinical diagnosis of opioid dependence
* Fluent in English or Spanish
* 18 years or older

Exclusion Criteria:

* Liver function tests (transaminase only) at five times or higher than normal level;
* Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) criteria for benzodiazepine abuse or dependence within the past 6 months;
* DSM-IV criteria for alcohol dependence within the past 6 months;
* Actively suicidal;
* Psychiatric impairment that impedes ability to consent (dementia, delusional, actively psychotic);
* Methadone dose exceeding levels allowing for safe transition to buprenorphine;
* Pregnant women and women actively trying to become pregnant;
* Clinical judgment of local site principal investigator that patient is inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Substance use outcomes measured by self-report | at 1, 3, 6, 9 and 12 months measured by self-report
Urine toxicology results | at 1, 3, 6, 9 and 12 months
Retention in and adherence to HIV care | at 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Quality of life | at 1, 3, 6, 9, and 12 months
HIV-related health outcomes | at 1, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University
Locations (1):
- Yale AIDS Program, New Haven, Connecticut, United States